CLINICAL TRIAL: NCT04754516
Title: Diagnosis of Short Stature in Children : Study of a Cohort of Small-sized Consulting Patients in 2017 and 2018
Brief Title: Diagnosis of Short Stature in Children : Study of a Cohort of Small-sized Consulting Patients
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0065
Record Dates: First submitted 2021-02-10; First posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Short Stature; Growth Delay
Keywords: Constitutional bone disease; Pediatrics
MeSH Terms: conditions — Dwarfism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Many patients consult in pediatric endocrinology because of their small size. In the majority of cases, this growth delays can be explained by a hormonal, gastroenterological cause, or a chronic disease.

Sometimes the reason for stunted growth can be constitutional bone disease, a genetic cause of short stature that is still underdiagnosed.

The investigators wish to describe and take stock of the various additional analyzes carried out and the various diagnoses made in patients who consulted in endocrino-pediatrics at the Montpellier University Hospital due to their short stature, in 2017 and 2018, in order to better screen patients with constitutional bone disease

ELIGIBILITY:
Inclusion criteria:

All the children who consulted for the first time because of their short stature, in pediatric endocrinology at the Montpellier University Hospital between January 2017 and December 2018

Exclusion criteria:

Patient already undergoing specialized medical follow-up due to his small size Major patient

Max Age: 17 Years | Healthy Volunteers: No
Age Groups: Child
Study Population: All the children who consulted for the first time because of their short stature, in pediatric endocrinology at the Montpellier University Hospital between January 2017 and December 2018
Sampling Method: Non-Probability Sample
Enrollment: 479 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-02-08 (Actual)

PRIMARY OUTCOMES:
Study the prevalence of different diagnoses of stature delay in children | 1 day
  Study the prevalence of different diagnoses of stature delay in children

CONTACTS AND LOCATIONS:
Overall Officials: Cyril Amouroux, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC